CLINICAL TRIAL: NCT00200889
Title: Auricular Vagal Nerve Stimulation for Gastric and Brain Outcomes
Brief Title: Mapping Auricular Vagus Nerve Circuitry
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Vitaly Napadow, Ph.D., Lic.Ac., Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2009P002177; 3OT2OD023867-01S2 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Acupuncture; Magnetic Resonance Imaging, Functional; Brain Mapping; healthy volunteers; Neuromodulation; gastric MRI

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to "Congruent" or "Incongruent" briefing groups. The Congruent group receives briefings including expectations of stimulation effects on gastric motility consistent with prior research in the literature. The Incongruent group receives briefings including expectations of stimulation effects on gastric motility inconsistent with prior research in the literature.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not made aware of the expectation manipulation nor their group assignment until the end of the final visit, at which point they are debriefed.
  Outcomes assessors will be blind to group assignments until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Congruent (Experimental): Participants receive briefings on expectations of stimulation effects on gastric motility consistent with the literature.
  Interventions: Device: active TEAS
- Incongruent (Experimental): Participants receive briefings on expectations of stimulation effects on gastric motility inconsistent with the literature.
  Interventions: Device: active TEAS

INTERVENTIONS:
Device: active TEAS — non-painful active transcutaneous electro-acupoint stimulation will be delivered to the abdomen and leg

SUMMARY:
This study will determine how noninvasive nerve stimulation affects human brain, stomach, and autonomic activity.

DETAILED DESCRIPTION:
Scientific research into the basic mechanisms underlying neuromodulation is relatively recent and incomplete. The purpose of the proposed study is to determine how a form of neuromodulation, transcutaneous electro-accupoint stimulation, which is non-invasive and non-painful, affects human brain, stomach, and autonomic activity. We will accomplish this by integrating whole brain functional MRI (fMRI) methodologies with gastric MRI and physiological monitoring.

This study will comprise 3 functional magnetic resonance imaging (fMRI) brain-gut scans, all while receiving the neuromodulation with varying parameters. Participants will also have their heart rate, breathing, and gastric activity monitored during all visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65
* Functional dyspepsia

Exclusion Criteria:

* Any condition contraindicating an fMRI brain scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain activity during functional magnetic resonance imaging (fMRI) | 1 hour
  Blood oxygen-level dependent (BOLD) signal change between active and inactive auricular tVNS
Stomach activity during gastric magnetic resonance imaging (MRI) | 30 minutes
  Gastric accommodation and sensitivity change between active and inactive auricular tVNS

SECONDARY OUTCOMES:
Electrogastrography (EGG) | 2 hours
  We will use EGG to measure slow wave myoelectrical activity, as measured by EGG power/peak frequency.
Electrocardiography (ECG) | 2 hours
  We will use ECG to examine high frequency heart rate variability (HF-HRV), i.e. the R-peak of the QRS complex.
Respiration | 2 hours
  Respiration will be measured in beats per minute (bpm).
Skin Conductance Levels (SCL) | 2 hours
  SCL will be measured in volts per second.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD, Principal Investigator — Harvard University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States